CLINICAL TRIAL: NCT00002844
Title: Bone Marrow Transplantation for Chronic Lymphocytic Leukemia
Brief Title: Bone Marrow Transplantation in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM90-106; P30CA016672 (NIH); MDA-DM-90106 (Other: UT MD Anderson Cancer Center); NCI-G96-1034; CDR0000065081 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-06-23 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; Cyclophosphamide; Cytoxan; Neosar; Bone Marrow Transplantation; total body irradiation; chronic lymphocytic leukemia; allogeneic; autologous
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; Stem Cell Transplantation; Whole-Body Irradiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclophosphamide + TBI + BMT (Experimental): TBI = Total Body Irradiation and BMT = Bone Marrow Transplantation (allogeneic or autologous bone marrow)
  Interventions: Drug: Cyclophosphamide; Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Autologous Bone Marrow Transplantation; Radiation: Total Body Irradiation (TBI)

INTERVENTIONS:
Drug: Cyclophosphamide — Daily intravenous infusions of cyclophosphamide for two days,
  Other Names: Cytoxan; Neosar
Procedure: Allogeneic Bone Marrow Transplantation — After completion of the TBI, allogeneic or autologous bone marrow infused intravenously.
  Other Names: Stem Cell Transplant
Procedure: Autologous Bone Marrow Transplantation — After completion of the TBI, allogeneic or autologous bone marrow infused intravenously.
  Other Names: Stem Cell Transplant
Radiation: Total Body Irradiation (TBI) — Following 2 days of cyclophosphamide, TBI in four daily exposures then bone marrow transplant.
  Other Names: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of bone marrow transplantation in treating patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: Examine the potential role for high dose cyclophosphamide, total body irradiation and bone marrow transplantation for patients with chronic lymphocytic leukemia who are at high risk for disease progression.

OUTLINE: Patients receive daily intravenous infusions of cyclophosphamide for two days, followed by total body irradiation in four daily exposures. After completion of the total body irradiation, allogeneic or autologous bone marrow is infused intravenously.

PROJECTED ACCRUAL: 50 patients are expected to be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Chronic lymphocytic leukemia (CLL) patients after initial relapse who have achieved a complete or partial remission with fludarabine therapy or after initial relapse or progression Prolymphocytic leukemia in first remission or after relapse Patients 15-65 years old who lack an HLA-identical sibling are eligible for autologous BM transplantation Patients 16-50 years old with an HLA identical or one antigen mismatched related donor are eligible for allogeneic BM transplantation

PATIENT CHARACTERISTICS: Age: 15-65 (See Disease Characteristics) Performance status: Zubrod no more than 2 Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: Cardiac ejection fraction at least 50% Pulmonary: DLCO at least 50% of predicted Other: No severe concomitant medical or psychiatric illnesses

PRIOR CONCURRENT THERAPY: No extensive prior radiotherapy which would prevent administration of total body radiation Patients may also participate in study MDA-DM-92082 for retroviral gene marking of the autologous marrow and blood cells

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 1991-03-05; Primary Completion 2002-06-05 (Actual); Study Completion 2002-06-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness of high dose cyclophosphamide, total body irradiation and bone marrow transplantation for chronic lymphocytic leukemia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org